CLINICAL TRIAL: NCT00560690
Title: Effect and Safety of Adding Metformin to the Standard Treatment of Hepatitis C on Sustained Viral Response
Brief Title: The Effect of Adding Metformin to the Treatment of Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shahin Merat, Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 83/53
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; metformin; Insulin Resistance
MeSH Terms: conditions — Hepatitis C; Insulin Resistance | interventions — Metformin; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): standard treatment with pegylated interferon and ribavirin + placebo
  Interventions: Drug: pegylated interferon; Drug: Ribavirin
- Metformin (Experimental): standard treatment with pegylated interferon and ribavirin + metformin
  Interventions: Drug: Metformin; Drug: pegylated interferon; Drug: Ribavirin

INTERVENTIONS:
Drug: Metformin — 500 mg oral three times a day for 6 months
  Arms: Metformin
Drug: pegylated interferon — 180 micrograms, or 1.5 micrograms/kg body weight weekly SQ injection for 6 or 12 months depending on genotype
Drug: Ribavirin — 800-1200 mg PO given in 2 divided doses for 6 to 12 months depending on weight and genotype

SUMMARY:
Insulin resistance is known to adversely effect viral response to treatment in hepatitis C patients

We are aiming to study the effect of an insulin sensitizer, metformin, in viral response of hepatitis C to treatment with pegylated interferon and ribavirin in a double blind randomized controlled trial

DETAILED DESCRIPTION:
Subjects with hepatitis C will be randomized to receive standard treatment with or without metformin. The results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis C
* Iranian nationality
* Treatment naive

Exclusion Criteria:

* cirrhosis
* diabetes mellitus
* HBV/HIV coinfection
* contraindications of metformin, interferon, ribavirin
* severe medical conditions (e.g. CHF, CRF, psychosis, ...)
* not consenting

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Sustained viral response, defined as undetectable virus RNA 6 months after end of treatment | 6 months after end of treatment

SECONDARY OUTCOMES:
adverse effects leading to discontinuation of treatment | anytime during the study
Rapid viral response, defined as undetectable viral RNA one month after start of treatment | one month after start of treatment
Early viral response, defined as undetectable viral RNA or 2 log drop in viral count three month after start of treatment | three months after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shahin Merat, MD, Principal Investigator — Digestive Disease Research Center, Medical Sciences / University of Tehran; Reza Malekzadeh, MD, Study Chair — Digestive Disease Research Center, Medical Sciences / University of Tehran
Locations (1):
- Shariati Hospital, Tehran, Tehran Province, Iran